CLINICAL TRIAL: NCT01077297
Title: Multicenter, Open-label, Non-comparative, Proof-of-concept, Phase 2a Study to Evaluate the Effect of a Single Infusion of Tezosentan on Pulmonary Vascular Resistance in Patients With Stable, Chronic Pulmonary Arterial Hypertension, Currently Not Treated With Endothelin Receptor Antagonists, Phosphodiesterase-5 Inhibitors or Prostacyclines
Brief Title: Tezosentan in Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment, the study was prematurely discontinued
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-051-206
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — tezosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tezosentan (Experimental)
  Interventions: Drug: Tezosentan

INTERVENTIONS:
Drug: Tezosentan — single infusion of tezosentan 5mg/h over 30 min corresponding to 2.5 mg

SUMMARY:
Multicenter, Open-label, Non-comparative, Proof-of-concept, Phase 2a Study to Evaluate the Effect of a Single Infusion of Tezosentan on Pulmonary Vascular Resistance in Patients With Stable, Chronic Pulmonary Arterial Hypertension, Currently Not Treated With Endothelin Receptor Antagonists, Phosphodiesterase-5 Inhibitors or Prostacyclines

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male and female patients 18 years of age or older
3. Patients with PAH according to one of the following subgroups of the Venice Classification Group 1:

   * Idiopathic (iPAH), or
   * Familial/heritable (FPAH), or
   * Associated (APAH) with collagen vascular disease
4. Modified NYHA functional class II-III
5. Documented hemodynamic diagnosis of PAH by right heart catheterization at Baseline:

   * Resting mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg and
   * Resting mean PVR ≥ 240 dyn•s•cm-5 and
   * Pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg

Exclusion Criteria:

1. Patients with PAH in Venice Classification Groups 2-5, and PAH Group 1 subgroups not covered by inclusion criterion no. 3
2. Hypotensive patients (systemic systolic blood pressure < 100 mmHg)
3. Patients with body weight < 50 kg (110 lbs)
4. Patients with moderate or severe hepatic impairment (Child-Pugh B and C)
5. Patients with clinically significant chronic renal insufficiency (serum creatinine > 2.5mg/dL / 221µmol/L)
6. Patients who have received any endothelin receptor antagonist (ERA) and/or any phosphodiesterase-5 (PDE-5) inhibitor within 28 days of Baseline
7. Patients who have received prostacyclin (epoprostenol) or prostacyclin analogs (e.g., treprostinil, iloprost) within 28 days of Baseline
8. Patients who have received any investigational drugs within 28 days of Baseline
9. Patients who have received cyclosporine A or tacrolimus within 28 days of Baseline
10. Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with the study
11. Life expectancy less than 12 months
12. Females who are lactating or pregnant or females who are not using a reliable method of birth control (failure rate less than 1% per year) during the study and for at least one month after study drug intake
13. Known hypersensitivity to any of the excipients of the drug formulation
14. Patients with positive response to vasoreactivity test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in PVR from Baseline to 30 minutes expresses as percent of the Baseline value. | 30 minutes

SECONDARY OUTCOMES:
Change in mean right arterial pressure (mRAP) from Baseline to 30 minutes | 30 minutes
Change in mPAP from Baseline to 30 min | 30 minutes
Change in total pulmonary resistance (TPR) from Baseline to 30 min | 30 minutes
Change in PCWP from Baseline to 30 min | 30 minutes
Change in cardiac output (CO) from Baseline to 30 min | 30 minutes
Change in cardiac index (CI) from Baseline to 30 min | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Lindberg, MD, Study Director — Actelion
Locations (5):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Baylor College of Medicine, Houston, Texas
- Hopital Antoine Béclère, Paris, Clamart, France
- Switzerland (2):
  - University Hospital of Basel, Clinic of Pneumology, Basel
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne